CLINICAL TRIAL: NCT05876208
Title: Measuring the Effectiveness of BAND Connect's VirtuaCare™ Asynchronous Telerehabilitation Platform in Increasing Patient Adherence for Total Shoulder Arthroplasty and Rotator Cuff Repair Physical Therapy Rehabilitatio
Brief Title: Increased Home-based Physical Therapy Adherence Using BAND Connect's VirtuaCare™ Platform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Brian Grawe, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM22053
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Injuries
Keywords: Rotator Cuff Repair; Anatomic and Reverse Total Shoulder
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will be using the BAND CVCP both in the clinic and at home to supplement the treatment protocols used in the clinic today.
  Interventions: Other: BAND Connect's VirtuaCare™ platform
- Group 2 (Placebo Comparator): Group 2 will receive standard-of-care physical therapy without the use of the BAND CVCP.
  Interventions: Other: Standard of Care Physical Therapy

INTERVENTIONS:
Other: BAND Connect's VirtuaCare™ platform — Band Connect provides a medical-grade and condition-specific platform that augments the clinician workflow by extending the in-clinic MSK rehabilitation experience into the patient's home - leading to higher quality personalized treatment and increased adherence with enhanced economics and reimbursement for the clinic.
  Arms: Group 1
Other: Standard of Care Physical Therapy — Standard of care physical therapy without the use of the BAND CVCP
  Arms: Group 2

SUMMARY:
This study aims to enhance at-home therapy by introducing a new device called the BAND Connect's VirtuaCare™ platform. The study aims to determine whether patients can improve their adherence to at-home exercises using this device. Currently, research indicates that only 35% of patients undergoing physical therapy treatment fully comply with their prescribed plans of care, often neglecting their at-home exercises. To address this issue, a set of smart exercise tools called VirtuaCare™ has been developed. This platform provides patients with instructions on performing at-home exercises and offers real-time biofeedback to help them adjust their form if necessary. The study seeks to evaluate the effectiveness of BAND CVCP in assisting patients and improving their overall success with at-home therapy.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of the BAND CVCP device with the standard physical therapy regimens provided by UC Health Orthopaedic Surgery. Participants undergoing shoulder surgeries performed by Dr. Brian Grawe will be randomly assigned to one of two groups. Group 1 will utilize the BAND CVCP both in the clinic and at home as a supplement to their treatment protocols. Group 2 will receive standard physical therapy without the BAND CVCP.

In Group 1, participants will be given access to the BAND CVCP and necessary materials during their first physical therapy appointment. The physical therapist will guide them through exercises using the device, recording their actions and providing real-time feedback. The BAND CVCP app on their provided Android phone will offer instructions for each exercise, eliminating the need to memorize the routine.

During clinic visits, Group 1 participants' progress will be reviewed using the BAND CVCP participant report. The report will display information such as completed exercises, form, pace, range of motion, and exertion, which is measured by sensors in the BAND CVCP handles. The therapist will help participants understand any corrections needed for their at-home exercises and make adjustments to their rehabilitation plan accordingly.

Both Group 1 and Group 2 participants will complete patient report outcomes at different intervals, including pre-operative scores, weekly visual analog scale assessments, and monthly assessments such as the Upper Extremity Functional Index (UEFI) or Quick Disabilities of Arm, Shoulder, and Hand (QuickDASH). Group 1 participants will complete these forms using the BAND CVCP's phone application, while Group 2 participants will use paper copies at the clinic.

Additional assessments will be conducted at the 3-month, 6-month, and discharge from care visits, which include the ASES, SST, and EQ-5D-5L forms. Group 1 participants will complete these assessments on the BAND CVCP's phone application, while Group 2 participants will use paper copies at the clinic.

This study aims to evaluate the effectiveness of the BAND CVCP device compared to standard physical therapy regimens and track participant rehabilitation outcomes throughout the process.

ELIGIBILITY:
Inclusion Criteria:

* Dr. Brian Grawe will perform surgery, and participants will be undergoing post-operative physical therapy rehabilitation at UC Health.
* Primary total shoulder arthroplasty and primary reverse total shoulder arthroplasty or Primary rotator cuff repair
* Outpatient physical therapy prescribed by the doctor for post-operative rehabilitation

Exclusion Criteria:

* Unplanned surgical procedure
* Partial shoulder replacement or revision shoulder replacement
* Revision rotator cuff repair
* Fracture surgeries
* Prior surgery within the last 5 years or less than 6 months between surgery on opposite shoulder
* Length of stay in hospital greater than 3 days
* Comorbidity: Uncontrolled diabetes patients; Diagnosed with cancer in the past 5 years or active disease; Any comorbidity that may impact compliance with the study protocol (completion of standard physical therapy rehabilitation procedures)
* Injuries related to workers' compensation
* Injuries involved in any pending litigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Visits | 12 weeks
  Number of visits with physical therapist

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Grawe, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuff DJ, Pupello DR. Prospective randomized study of arthroscopic rotator cuff repair using an early versus delayed postoperative physical therapy protocol. J Shoulder Elbow Surg. 2012 Nov;21(11):1450-5. doi: 10.1016/j.jse.2012.01.025. Epub 2012 May 2. PMID 22554876
- [Background] Dahl-Popolizio S, Loman J, Cordes CC. Comparing Outcomes of Kinect Videogame-Based Occupational/Physical Therapy Versus Usual Care. Games Health J. 2014 Jun;3(3):157-61. doi: 10.1089/g4h.2014.0002. Epub 2014 Apr 17. PMID 26196174
- [Background] Keener JD, Galatz LM, Stobbs-Cucchi G, Patton R, Yamaguchi K. Rehabilitation following arthroscopic rotator cuff repair: a prospective randomized trial of immobilization compared with early motion. J Bone Joint Surg Am. 2014 Jan 1;96(1):11-9. doi: 10.2106/JBJS.M.00034. PMID 24382719
- [Background] Palazzo C, Klinger E, Dorner V, Kadri A, Thierry O, Boumenir Y, Martin W, Poiraudeau S, Ville I. Barriers to home-based exercise program adherence with chronic low back pain: Patient expectations regarding new technologies. Ann Phys Rehabil Med. 2016 Apr;59(2):107-13. doi: 10.1016/j.rehab.2016.01.009. Epub 2016 Apr 1. PMID 27050664
- [Background] Raaben M, Holtslag HR, Leenen LPH, Augustine R, Blokhuis TJ. Real-time visual biofeedback during weight bearing improves therapy compliance in patients following lower extremity fractures. Gait Posture. 2018 Jan;59:206-210. doi: 10.1016/j.gaitpost.2017.10.022. Epub 2017 Oct 20. PMID 29078134
- [Background] Sluijs EM, Kok GJ, van der Zee J. Correlates of exercise compliance in physical therapy. Phys Ther. 1993 Nov;73(11):771-82; discussion 783-6. doi: 10.1093/ptj/73.11.771. PMID 8234458
- [Background] Arndt J, Clavert P, Mielcarek P, Bouchaib J, Meyer N, Kempf JF; French Society for Shoulder & Elbow (SOFEC). Immediate passive motion versus immobilization after endoscopic supraspinatus tendon repair: a prospective randomized study. Orthop Traumatol Surg Res. 2012 Oct;98(6 Suppl):S131-8. doi: 10.1016/j.otsr.2012.05.003. Epub 2012 Sep 1. PMID 22944392
- [Background] Denard PJ, Ladermann A, Burkhart SS. Prevention and management of stiffness after arthroscopic rotator cuff repair: systematic review and implications for rotator cuff healing. Arthroscopy. 2011 Jun;27(6):842-8. doi: 10.1016/j.arthro.2011.01.013. PMID 21624680
- [Background] Huberty DP, Schoolfield JD, Brady PC, Vadala AP, Arrigoni P, Burkhart SS. Incidence and treatment of postoperative stiffness following arthroscopic rotator cuff repair. Arthroscopy. 2009 Aug;25(8):880-90. doi: 10.1016/j.arthro.2009.01.018. PMID 19664508
- [Background] Koo SS, Parsley BK, Burkhart SS, Schoolfield JD. Reduction of postoperative stiffness after arthroscopic rotator cuff repair: results of a customized physical therapy regimen based on risk factors for stiffness. Arthroscopy. 2011 Feb;27(2):155-60. doi: 10.1016/j.arthro.2010.07.007. Epub 2010 Oct 20. PMID 20970299
- [Background] Carbonaro N, Lucchesi I, Lorusssi F, Tognetti A. Tele-monitoring and tele-rehabilitation of the shoulder muscular-skeletal diseases through wearable systems. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:4410-4413. doi: 10.1109/EMBC.2018.8513371. PMID 30441330
- [Background] Brandao AF, Dias DR, Castellano G, Parizotto NA, Trevelin LC. RehabGesture: An Alternative Tool for Measuring Human Movement. Telemed J E Health. 2016 Jul;22(7):584-9. doi: 10.1089/tmj.2015.0139. Epub 2016 May 12. PMID 27172389
- [Background] Kennedy JS, Garrigues GE, Pozzi F, Zens MJ, Gaunt B, Phillips B, Bakshi A, Tate AR. The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation for anatomic total shoulder arthroplasty. J Shoulder Elbow Surg. 2020 Oct;29(10):2149-2162. doi: 10.1016/j.jse.2020.05.019. Epub 2020 Jun 10. PMID 32534209
- [Background] Brameier DT, Hirscht A, Kowalsky MS, Sethi PM. Rehabilitation Strategies After Shoulder Arthroplasty in Young and Active Patients. Clin Sports Med. 2018 Oct;37(4):569-583. doi: 10.1016/j.csm.2018.05.007. PMID 30201171
- [Background] Ikard ST Jr, Farmer KW, Struk AM, Garvan CS, Gillespy A, Wright TW. Rotator Cuff Dysfunction after Anatomic Total Shoulder Arthroplasty: Who is at Risk? J Surg Orthop Adv. 2020 Spring;29(1):31-35. PMID 32223863